CLINICAL TRIAL: NCT02248597
Title: Haploidentical Stem Cell Transplant Using Post Transplant Cyclophosphamide for GvHD Prophylaxis: A Pilot Study
Brief Title: Donor Stem Cell Transplant Followed by Cyclophosphamide in Treating Patients With Hematological Diseases
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00029210; NCI-2014-01898 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CCCWFU 97214 (Other: Comprehensive Cancer Center of Wake Forest University); P30CA012197 (NIH)
Record Dates: First submitted 2014-09-23; First posted 2014-09-25 (Estimated); Results first posted 2023-10-11 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Graft Versus Host Disease; Hematopoietic/Lymphoid Cancer
MeSH Terms: conditions — Graft vs Host Disease; Hematologic Neoplasms | interventions — fludarabine phosphate; Busulfan; Cyclophosphamide; Tacrolimus; Mycophenolic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (stem cell transplant with GVHD prophylaxis) (Experimental): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV QD on days -6 to -2. Patients receiving myeloablative conditioning receive busulfan IV every 6 hours for 16 doses on days -7 to -4 and patients receiving reduced intensity conditioning receive busulfan IV every 6 hours for 8 doses on days -5 to -4. Patients also receive cyclophosphamide IV QD on days -3 and -2
  TRANSPLANT: Patients undergo stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide QD on days 3 and 4, tacrolimus on days 5-180, and mycophenolate mofetil on days 5-35. Allogeneic hematopoietic stem cell transplantation
  Interventions: Drug: fludarabine phosphate; Drug: busulfan; Drug: cyclophosphamide; Procedure: allogeneic hematopoietic stem cell transplantation; Drug: tacrolimus; Drug: mycophenolate mofetil

INTERVENTIONS:
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: busulfan — Given IV
  Other Names: BSF; BU; Misulfan; Mitosan; Myeloleukon
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Procedure: allogeneic hematopoietic stem cell transplantation — Undergo myeloablative or reduced intensity allogeneic stem cell transplant
Drug: tacrolimus
  Other Names: FK 506; Prograf
Drug: mycophenolate mofetil
  Other Names: Cellcept; MMF

SUMMARY:
This pilot clinical trial studies donor stem cell transplant followed by cyclophosphamide in treating patients with hematological diseases. Giving chemotherapy before a donor stem cell transplant helps stop the growth of cells in the bone marrow, including normal blood-forming cells (stem cells) and cancer cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells (called graft-versus-host disease). Giving cyclophosphamide after the transplant may stop this from happening.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if haploidentical stem cell transplant using post-transplant cyclophosphamide results in 60% or better disease free survival (DFS) at 12 months at our institution.

SECONDARY OBJECTIVES:

I. To determine the rate of acute and chronic graft-versus-host disease (GvHD), non-relapse mortality, and relapse.

OUTLINE:

PREPARATIVE REGIMEN: Patients receive fludarabine phosphate intravenously (IV) once daily (QD) on days -6 to -2. Patients receiving myeloablative conditioning receive busulfan IV every 6 hours for 16 doses on days -7 to -4 and patients receiving reduced intensity conditioning receive busulfan IV every 6 hours for 8 doses on days -5 to -4. Patients also receive cyclophosphamide IV QD on days -3 and -2

TRANSPLANT: Patients undergo stem cell transplant on day 0.

GVHD PROPHYLAXIS: Patients receive cyclophosphamide QD on days 3 and 4, tacrolimus on days 5-180, and mycophenolate mofetil on days 5-35.

After completion of study treatment, patients are followed up periodically for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of a hematological malignancy requiring an allogeneic stem cell transplant consistent with the standard of care
* Remission of any acute hematologic malignancy or adequate disease control for chronic malignancies.
* Ages 18-69 years old.
* Available familial haploidentical (4 to 6 out of 8 HLA loci-matched) donor

Exclusion Criteria:

* Significant organ dysfunction defined as: LV EF < 50% (evaluated by echocardiogram or MRI), DLCO or FEV1 < 65% predicted, AST/ALT > 2.5 x ULN, Bilirubin > 1.5 x ULN, Serum creatinine > 2mg/dL, dialysis, or prior renal transplant
* HIV positive (Recipients who are positive for hepatitis B (HBV), hepatitis C (HCV) or human T-cell lymphotropic virus (HTLV-I/II) are not excluded from participation)
* Positive pregnancy test for women of childbearing age.
* Major anticipated illness or organ failure incompatible with survival form transplant.
* Severe psychiatric illness or mental deficiency sufficiently severe as to make compliance with the transplant treatment unlikely and informed consent impossible.

Ages: 18 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2015-02-25 (Actual); Primary Completion 2022-01-18 (Actual); Study Completion 2023-01-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dianna S. Howard, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Comprehensive Cancer Center of Wake Forest University, Winston-Salem, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (Stem Cell Transplant With GVHD Prophylaxis): PREPARATIVE REGIMEN: Patients receive fludarabine phosphate IV QD on days -6 to -2. Patients receiving myeloablative conditioning receive busulfan IV every 6 hours for 16 doses on days -7 to -4 and patients receiving reduced intensity conditioning receive busulfan IV every 6 hours for 8 doses on days -5 to -4. Patients also receive cyclophosphamide IV QD on days -3 and -2
  TRANSPLANT: Patients undergo stem cell transplant on day 0.
  GVHD PROPHYLAXIS: Patients receive cyclophosphamide QD on days 3 and 4, tacrolimus on days 5-180, and mycophenolate mofetil on days 5-35. Allogeneic hematopoietic stem cell transplantation
  fludarabine phosphate: Given IV
  busulfan: Given IV
  cyclophosphamide: Given IV
  allogeneic hematopoietic stem cell transplantation: Undergo myeloablative or reduced intensity allogeneic stem cell transplant
  tacrolimus
  mycophenolate mofetil
Period: Overall Study
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Started | 27
Completed | 27
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
Age, Continuous [Mean (Standard Deviation); unit: years] — Participants were 18-69 years
  years | 53.4 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12
  Male | 15
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 18
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Number; unit: participants]
  United States | 27

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Disease Free Survival Probability
Description: The percentage of patients who experience death or disease relapse by one year will be calculated and a corresponding 95% confidence interval will be constructed using the normal approximation for binomial proportions. The survival function will be estimated and plotted using the method of Kaplan and Meier.
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
percentage of participants | 51.8 [33.0 to 70.7]

2. Secondary Outcome: Rate of Acute GvHD
Description: Kaplan-Meier estimation of the rate of acute GvHD in the study population at one year with a 95% confidence interval.
Time Frame: 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
percentage of participants | 51.8 [30.0 to 70.7]

3. Secondary Outcome: Overall Survival
Description: The survival function will be estimated and plotted using the method of Kaplan and Meier.
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
percentage of participants | 66.7 [45.7 to 81.1]

4. Secondary Outcome: Progression Free Survival
Description: Kaplan-Meier estimation of the percentage of patients who are alive without progressive disease at one year.
Time Frame: At 12 months
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
percentage of participants | 51.8 [31.9 to 68.5]

5. Secondary Outcome: Relapse-free Mortality
Description: Non-relapse mortality will be defined as time from registration to death due to anything other than relapse of hematological malignancy. Patients who relapse will be treated as a competing risk.
Time Frame: At 12 months
Measure: Mean (95% Confidence Interval); unit: days
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
Number analyzed (Participants) | 27
days | 86.8 [63.4 to 95.7]

ADVERSE EVENTS:
Time Frame: Adverse events were monitored 100 days post-transplant. Deaths were assessed for 1 year.
Arm/Group | Treatment (Stem Cell Transplant With GVHD Prophylaxis)
All-Cause Mortality (participants affected / at risk) | 13/27
Serious Adverse Events (participants affected / at risk) | 27/27
Other Adverse Events (participants affected / at risk) | 27/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Stem Cell Transplant With GVHD Prophylaxis) (N=27)
Death (General disorders) | 3 (3)
Anemia (Blood and lymphatic system disorders) | 8 (8)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 2 (2)
Lymphocyte count decreased (Investigations) | 20 (20)
Neutrophil count decreased (Investigations) | 15 (15)
Platelet count decreased (Investigations) | 23 (23)
White blood cell count decreased (Investigations) | 24 (24)
Retinal vascular disorder (Eye disorders) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Fever (General disorders) | 1 (1)
Ongoing viremia (Infections and infestations) | 1 (1)
Stenotrophomonas (Infections and infestations) | 1 (1)
Kidney infection (Infections and infestations) | 1 (1)
Lung infection (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Chronic kidney disease (Renal and urinary disorders) | 3 (3)
Hematuria (Renal and urinary disorders) | 1 (1)
Renal hemorrhage (Renal and urinary disorders) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hypotension (Vascular disorders) | 1 (1)
Lymphedema (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Stem Cell Transplant With GVHD Prophylaxis) (N=27)
Anemia (Blood and lymphatic system disorders) | 24 (24)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 2 (2)
ALC decrease (Blood and lymphatic system disorders) | 2 (2)
Pancytopenia (Blood and lymphatic system disorders) | 2 (2)
Activated partial thromboplastin time prolonged (Investigations) | 6 (6)
Alanine aminotransferase increased (Investigations) | 7 (7)
Alkaline phosphatase increased (Investigations) | 5 (5)
Aspartate aminotransferase increased (Investigations) | 5 (5)
Bilirubin increased (Investigations) | 9 (9)
Cardiac troponin I increased (Investigations) | 2 (2)
Creatinine increased (Investigations) | 7 (7)
Lymphocyte count decreased (Investigations) | 16 (16)
Neutrophil count decreased (Investigations) | 13 (13)
Platelet count decreased (Investigations) | 19 (19)
White blood cell count decreased (Investigations) | 17 (17)
Hypervolemia (Cardiac disorders) | 2 (2)
Heart failure (Cardiac disorders) | 2 (2)
Palpitations (Cardiac disorders) | 2 (2)
Periocardial effusions (Cardiac disorders) | 3 (3)
Sinus bradycardia (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 14 (14)
Fatigue (General disorders) | 22 (22) — Asthenia, lethargy, malaise
Dry eye (Eye disorders) | 3 (3)
Abdominal distension (Gastrointestinal disorders) | 5 (5)
Abdominal pain (Gastrointestinal disorders) | 12 (12)
Anal pain (Gastrointestinal disorders) | 4 (4)
Ascites (Gastrointestinal disorders) | 2 (2)
Bloating (Gastrointestinal disorders) | 2 (2)
Constipation (Gastrointestinal disorders) | 5 (5)
Diarrhea (Gastrointestinal disorders) | 21 (21)
Dry mouth (Gastrointestinal disorders) | 10 (10)
Dysphagia (Gastrointestinal disorders) | 4 (4)
Esophagitis (Gastrointestinal disorders) | 4 (4)
Flatulence (Gastrointestinal disorders) | 2 (2)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 4 (4)
Hemorrhoids (Gastrointestinal disorders) | 4 (4)
Oral mucositis (Gastrointestinal disorders) | 11 (11)
Nausea (Gastrointestinal disorders) | 21 (21)
Oral hemorrhage (Gastrointestinal disorders) | 2 (2)
Oral pain (Gastrointestinal disorders) | 5 (5)
Dysgeusia (Nervous system disorders) | 11 (11)
Vomiting (Gastrointestinal disorders) | 11 (11)
Chills (General disorders) | 13 (13)
Edema, face (General disorders) | 3 (3)
Edema, limbs (General disorders) | 14 (14)
Gait disturbance (General disorders) | 3 (3)
Hypothermia (General disorders) | 2 (2)
Infusion related reaction (General disorders) | 3 (3)
Localized edema (General disorders) | 3 (3)
Malaise (General disorders) | 3 (3)
Non-cardiac chest pain (General disorders) | 5 (5)
Pain (General disorders) | 8 (8)
Cytokine release syndrome (Immune system disorders) | 4 (4)
Catheter related infection (Infections and infestations) | 4 (4)
BK viruria urine (Infections and infestations) | 4 (4)
CMV Miremia (Investigations) | 2 (2)
Lung infection (Infections and infestations) | 7 (7)
Mucosal infection (Infections and infestations) | 2 (2)
Papulopustular rash (Infections and infestations) | 2 (2)
Skin infection (Infections and infestations) | 3 (3)
Urinary tract infection (Infections and infestations) | 5 (5)
Bruising (Injury, poisoning and procedural complications) | 3 (3)
Fall (Injury, poisoning and procedural complications) | 2 (2)
Electrocardiogram QT corrected interval prolonged (Investigations) | 6 (6)
Weight gain (Investigations) | 8 (8)
Weight loss (Investigations) | 9 (9)
Alkalosis (Metabolism and nutrition disorders) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 15 (15)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (16)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (3)
Hypermagnesemia (Metabolism and nutrition disorders) | 2 (2)
Hypernatremia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 15 (15)
Hypocalcemia (Metabolism and nutrition disorders) | 12 (12)
Hypoglycemia (Metabolism and nutrition disorders) | 7 (7)
Hypokalemia (Metabolism and nutrition disorders) | 15 (15)
Hypomagnesemia (Metabolism and nutrition disorders) | 16 (16)
Hyponatremia (Metabolism and nutrition disorders) | 14 (14)
Hypophosphatemia (Metabolism and nutrition disorders) | 6 (6)
Malnutrition (Metabolism and nutrition disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 10 (10)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 12 (12)
Myalgia (Musculoskeletal and connective tissue disorders) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 10 (10)
Dizziness (Nervous system disorders) | 9 (9)
Encephalopathy (Nervous system disorders) | 2 (2)
Headache (Nervous system disorders) | 16 (16)
Lethargy (Nervous system disorders) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 2 (2)
Presyncope (Nervous system disorders) | 5 (5)
Somnolence (Nervous system disorders) | 2 (2)
Tremor (Nervous system disorders) | 3 (3)
Anxiety (Psychiatric disorders) | 3 (3)
Confusion (Psychiatric disorders) | 5 (5)
Depression (Psychiatric disorders) | 5 (5)
Insomnia (Psychiatric disorders) | 6 (6)
Bladder spasm (Renal and urinary disorders) | 3 (3)
Proteinuria (Renal and urinary disorders) | 5 (5)
Urinary frequency (Renal and urinary disorders) | 7 (7)
Urinary retention (Renal and urinary disorders) | 4 (4)
Urinary tract pain (Renal and urinary disorders) | 7 (7)
Urinary urgency (Renal and urinary disorders) | 2 (2)
Scrotal pain (Reproductive system and breast disorders) | 3 (3)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 14 (14)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (5)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 7 (7)
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 12 (12)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 2 (2)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 2 (2)
Dry skin (Skin and subcutaneous tissue disorders) | 7 (7)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 4 (4)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (8)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 12 (12)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (2)
SKin hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 (2)
Skin ulceration (Skin and subcutaneous tissue disorders) | 5 (5)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2)
Flushing (Vascular disorders) | 2 (2)
Hematoma (Vascular disorders) | 2 (2)
Hot flashes (Vascular disorders) | 4 (4)
Hypertension (Vascular disorders) | 9 (9)
Hypotension (Vascular disorders) | 10 (10)
Febrile neutropenia (Blood and lymphatic system disorders) | 11 (11)
Fever (General disorders) | 18 (18)
Acute kidney injury (Renal and urinary disorders) | 6 (6)
Chronic kidney disease (Renal and urinary disorders) | 8 (8)
Hematuria (Renal and urinary disorders) | 7 (7)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-03-12): https://cdn.clinicaltrials.gov/large-docs/97/NCT02248597/Prot_SAP_001.pdf
  • Informed Consent Form (2021-02-22): https://cdn.clinicaltrials.gov/large-docs/97/NCT02248597/ICF_000.pdf